CLINICAL TRIAL: NCT03544645
Title: Are Audiovisual Educational Materials Superior to Printed Educational Materials in Improving Insulin Awareness Among Saudi Type 2 Diabetic Patients in Primary Care Setting?
Brief Title: Are Audiovisual Materials Superior to Printed Materials in Improving Awareness Among Type 2 Diabetic Patients?
Acronym: SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Mohammad Alsaif, bachelor degree in medicine, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KingAbdullahIMRC
Record Dates: First submitted 2018-04-30; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic Education; audiovisual material; Manual material
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): This group received a printed material "brochure" as an educational material
  Interventions: Other: Printed material "brochure"
- intervention group (Experimental): This group received an audiovisual material "video" as an educational material
  Interventions: Other: Audiovisual material "video"

INTERVENTIONS:
Other: Audiovisual material "video" — an educational video which has content of knowledge, attitude, behavior, and barriers towards insulin therapy.
  Arms: intervention group
Other: Printed material "brochure" — an educational brochure which has content of knowledge, attitude, behavior, and barriers towards insulin theray.
  Arms: control group

SUMMARY:
This research evaluates the effectiveness of video educations against patients fixed believes and knowledge that either not precise or overestimated, and compare with classic educational method such as Brochure. As many researches indicates the difficulties to initiate insulin therapy for type 2 diabetic patients due to overestimated barriers such as needle anxiety, feelings of guilt and failure, concerns about hypoglycemia, sense of loss of control over one's life and reduced quality of life. This research will introduce different educational tools to evaluate their effectiveness in breaking psychological insulin barriers.

DETAILED DESCRIPTION:
Introduction This research evaluates the effectiveness of video educations against patients fixed believes and knowledge that either not precise or overestimated, and compare with classic educational method such as Brochure. As many researches indicates the difficulties to initiate insulin therapy for type 2 diabetic patients due to overestimated barriers such as needle anxiety, feelings of guilt and failure, concerns about hypoglycemia, sense of loss of control over one's life and reduced quality of life. This research will introduce different educational tools to evaluate their effectiveness in breaking psychological insulin barriers.

Methodology It's a randomized controlled trial. Validated questionnaire (ITAS) was used to evaluate the psychological insulin barriers, video and Brochures were devolved as educational materials contain same contents and validated. Study conducted in King Abdulaziz city housing with total sample size of 126. They were divided into intervention group (video group) and controlled group (Brochure group). Both group filled the same questionnaire before the intervention. And then immediately after the intervention. Six weeks later, both groups filled the same questionnaire to measure the long-term effects.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients
2. Age group from 30 to 70 years
3. A1c = 8 mg/dL or above
4. Both genders

Exclusion Criteria:

1. Pregnant women
2. Blindness or profound vision loss
3. Severe mental problems e.g. Psychosis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
compare the impact of audiovisual educational materials verses printed educational materials | 6 weeks
  compare intervention versus control on type 2 diabetic patients' knowledge, attitude and practice towards insulin therapy by assessing the patients before, directly after and 6 weeks after the intervention using a validated questionnaire (ITAS) to evaluate the psychological insulin barriers, both intervention and control were devolved as educational materials contain same contents and validated

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud bin Abdulaziz University for Health Sciences, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided